CLINICAL TRIAL: NCT05485636
Title: Degenerative Lumbar Scoliosis: a Multi-center Study
Brief Title: Degenerative Lumbar Scoliosis
Acronym: DLS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Hebei Medical University Third Hospital (Other); Tianjin Hospital (Other); West China Hospital (Other); Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Nanchang University (Other); Henan Provincial People's Hospital (Other); The First People's Hospital of Yunnan (Other)
Responsible Party: Sponsor
Other Study IDs: M2022381
Record Dates: First submitted 2022-07-04; First posted 2022-08-03 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-07

CONDITIONS: Degenerative Scoliosis; Scoliosis Lumbar Region
Keywords: degenerative, lumbar, scoliosis, outcome
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- degenerative lumbar scoliosis postoperative group: This group contains patients who have undergone spinal surgery for degenerative lumbar scoliosis.
  No interventions are designed to be administered.

SUMMARY:
This is a retrospective, observational multi-center study. The participants undergone lumbar spine surgery for degenerative lumbar scoliosis and followed up for at least 2 years are retrospectively enrolled from 8 centers. This study mainly focuses on the short-term and long-term outcomes of lumbar surgery in participants with degenerative lumbar scoliosis, and that how much the surgical outcomes are related with demographic, surgical, and radiographic features before and after surgery. The objective is to offer more detailed clinical evidence to guide the surgical strategy development for degenerative lumbar scoliosis.

DETAILED DESCRIPTION:
Degenerative lumbar scoliosis is a spinal deformity that typically develops among adults over 50 years old. Characterized with low back pain, leg pain and abnormal body posture to various degrees, patients are mostly offered conservative treatment in early stages, and then resort to surgical treatment when medication fail to achieve alleviation. The surgical procedures to treat degenerative lumbar scoliosis include spinal decompression, fusion, and instrumentation, or a combination of several of the above. Osteotomy is generally required when it comes to rigid deformity. However, surgical treatment strategies are complicated by factors comprising osteoporosis, paraspinal muscle degeneration, common yet severe postoperative complications resulting from specific surgical methods, and chronic metabolic diseases and so on. A detailed and individualized surgical planning has been under debate and development continuously. Also, most previous classifications and researches are centered on the population of the white. Representative data of the yellow people, especially Chinese people, from multicentric studies are scarce.

Patients undergone surgeries for degenerative lumbar scoliosis in 8 hospitals in China between 2010 and 2020 are retrospectively selected and enrolled. Patients' clinical data from pre-operation, post-operation and the last follow-up are revaluated. General patient data are collected after informed consent, such as age, gender, height, weight, body mass index and bone mineral density measured in T-scores, together with surgical data including operation duration, blood loss, physical status grades based on the American Society of Anesthesiologists Classification, surgical approaches, upper instrumented vertebra, lowest instrumented vertebra, osteotomy grades based on Schwab Classification, osteotomy levels, lumbosacral curve levelling approaches, cemented vertebrae, and perioperative complications. Radiographic parameters of the spine are also measured from X-rays, including the upper end vertebra of the major curve, apical vertebral translation, Cobb angles of the major and fractional curves, coronal balance distance, coronal classification of the deformity based on the Drum Tower Classification, L4 and L5 tilt on the coronal plane, lumbar tilt, thoracic kyphosis, lumbar lordosis, thoracolumbar kyphosis, sagittal vertical axis, T1 pelvic angle, pelvic tilt, sacral slope, L4-S1 lordotic angle, and proximal junctional angle. Clinical outcomes assessed with Japanese Orthopaedic Association score, Oswestry Disability Index and visual analogue scale of leg/back pain are also gathered. Correlation between demographic, surgical, and radiographic parameters and clinical outcomes are statistically explored, in order to find indexes that help group and match patients with their optimum surgical strategies.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years old
* diagnosed with degenerative lumbar scoliosis with X-ray before surgery
* Cobb angle of the major curve ≥ 20°
* with signs and/or symptoms of low back pain and/or leg pain, torso imbalance, and spinal nerve compression
* followed up for at least 2 years after the surgery

Exclusion Criteria:

* scoliosis caused by infection, trauma or tumor.
* classified as adult idiopathic scoliosis, congenital scoliosis, and scoliosis caused by neuromuscular diseases
* previous history of spinal surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the orthopaedic department of the eight medical centers, patients undergone spinal surgery for degenerative lumbar scoliosis are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical complications | 24 months
  Mechanical complications at the last follow-up, including proximal junctional kyphosis, proximal junctional failure, distal junctional kyphosis, distal junctional failure, instrument breakage, pedicle screw loosening, pseudoarthrosis, and others.

SECONDARY OUTCOMES:
Radiological angular parameters | 3 months, 6 months, 12 months, 24 months
  Radiological angular parameters measured on anteroposterior and lateral radiographs, including: 1) major and lumbosacral Cobb angle, 2) L4, L5 and upper instrumented vertebra (UIV) tilt, 3)T1-UIV Cobb angle, 4) thoracic kyphosis, 5) lumbar lordosis, 6) thoracolumbar kyphosis, 7) T1 pelvic angle, 8) pelvic incidence, 9) pelvic tilt, 10) sacral slope, 11) lordosis tilt, 12) proximal junctional angle, and 13) L4-S1 lumbar lordosis.
Radiological distance parameters | 3 months, 6 months, 12 months, 24 months
  Radiological distance parameters measured on anteroposterior and lateral radiographs, including: 1) coronal balance distance, 2) sagittal vertical axis, 3) apical vertebral translation.
Back pain | 3 months, 6 months, 12 months, 24 months
  The Visual Analogue Scale (VAS 0-10) is adopted to evaluate back pain, with higher scores indicating severer pain.
Leg pain | 3 months, 6 months, 12 months, 24 months
  The Visual Analogue Scale (VAS 0-10) is adopted to evaluate leg pain, with higher scores indicating severer pain.
Disability | 3 months, 6 months, 12 months, 24 months
  The Japanese Orthopaedic Association (JOA 0-29) Scores is used to assess disability, with lower scores indicating severer disability. The Oswestry Disability Index (ODI 0-100%) is also used to assess disability, with higher percentages indicating severer disability.

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, M.D., Principal Investigator — Peking University Third Hospital
Locations (8):
- China (8):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
We will make the clinical study report available half a year after the publication of the results of the study.
Supporting Information: CSR
Time Frame: The IPD will become available half a year after the publication of the results of the study.
Access Criteria: The IPD is available to the readers of the journal in which our research is published. The corresponding author of the published papers will review the requests.

REFERENCES:
- [Background] Pritchett JW, Bortel DT. Degenerative symptomatic lumbar scoliosis. Spine (Phila Pa 1976). 1993 May;18(6):700-3. doi: 10.1097/00007632-199305000-00004. PMID 8516697
- [Background] Oskouian RJ Jr, Shaffrey CI. Degenerative lumbar scoliosis. Neurosurg Clin N Am. 2006 Jul;17(3):299-315, vii. doi: 10.1016/j.nec.2006.05.002. PMID 16876030
- [Background] Koerner JD, Reitman CA, Arnold PM, Rihn J. Degenerative Lumbar Scoliosis. JBJS Rev. 2015 Apr 7;3(4):e1. doi: 10.2106/JBJS.RVW.N.00061. No abstract available. PMID 27490255
- [Background] Xu L, Sun X, Huang S, Zhu Z, Qiao J, Zhu F, Mao S, Ding Y, Qiu Y. Degenerative lumbar scoliosis in Chinese Han population: prevalence and relationship to age, gender, bone mineral density, and body mass index. Eur Spine J. 2013 Jun;22(6):1326-31. doi: 10.1007/s00586-013-2678-8. Epub 2013 Jan 30. PMID 23361532
- [Background] Schwab F, Dubey A, Gamez L, El Fegoun AB, Hwang K, Pagala M, Farcy JP. Adult scoliosis: prevalence, SF-36, and nutritional parameters in an elderly volunteer population. Spine (Phila Pa 1976). 2005 May 1;30(9):1082-5. doi: 10.1097/01.brs.0000160842.43482.cd. PMID 15864163
- [Background] Jimbo S, Kobayashi T, Aono K, Atsuta Y, Matsuno T. Epidemiology of degenerative lumbar scoliosis: a community-based cohort study. Spine (Phila Pa 1976). 2012 Sep 15;37(20):1763-70. doi: 10.1097/BRS.0b013e3182575eaa. PMID 22487710
- [Background] Diebo B, Liu S, Lafage V, Schwab F. Osteotomies in the treatment of spinal deformities: indications, classification, and surgical planning. Eur J Orthop Surg Traumatol. 2014 Jul;24 Suppl 1:S11-20. doi: 10.1007/s00590-014-1471-7. Epub 2014 May 11. PMID 24816823
- [Background] Protopsaltis T, Schwab F, Bronsard N, Smith JS, Klineberg E, Mundis G, Ryan DJ, Hostin R, Hart R, Burton D, Ames C, Shaffrey C, Bess S, Errico T, Lafage V; International Spine Study Group. TheT1 pelvic angle, a novel radiographic measure of global sagittal deformity, accounts for both spinal inclination and pelvic tilt and correlates with health-related quality of life. J Bone Joint Surg Am. 2014 Oct 1;96(19):1631-40. doi: 10.2106/JBJS.M.01459. PMID 25274788
- [Background] Diebo BG, Oren JH, Challier V, Lafage R, Ferrero E, Liu S, Vira S, Spiegel MA, Harris BY, Liabaud B, Henry JK, Errico TJ, Schwab FJ, Lafage V. Global sagittal axis: a step toward full-body assessment of sagittal plane deformity in the human body. J Neurosurg Spine. 2016 Oct;25(4):494-499. doi: 10.3171/2016.2.SPINE151311. Epub 2016 May 20. PMID 27203811
- [Background] Bao H, Yan P, Qiu Y, Liu Z, Zhu F. Coronal imbalance in degenerative lumbar scoliosis: Prevalence and influence on surgical decision-making for spinal osteotomy. Bone Joint J. 2016 Sep;98-B(9):1227-33. doi: 10.1302/0301-620X.98B9.37273. PMID 27587525
- [Background] Wang H, Wang L, Sun Z, Jiang S, Li W. Posterior column osteotomy plus unilateral cage strutting for correction of lumbosacral fractional curve in degenerative lumbar scoliosis. J Orthop Surg Res. 2020 Oct 20;15(1):482. doi: 10.1186/s13018-020-02011-y. PMID 33081812
- [Background] Schwab FJ, Smith VA, Biserni M, Gamez L, Farcy JP, Pagala M. Adult scoliosis: a quantitative radiographic and clinical analysis. Spine (Phila Pa 1976). 2002 Feb 15;27(4):387-92. doi: 10.1097/00007632-200202150-00012. PMID 11840105
- [Background] Schwab FJ, Blondel B, Bess S, Hostin R, Shaffrey CI, Smith JS, Boachie-Adjei O, Burton DC, Akbarnia BA, Mundis GM, Ames CP, Kebaish K, Hart RA, Farcy JP, Lafage V; International Spine Study Group (ISSG). Radiographical spinopelvic parameters and disability in the setting of adult spinal deformity: a prospective multicenter analysis. Spine (Phila Pa 1976). 2013 Jun 1;38(13):E803-12. doi: 10.1097/BRS.0b013e318292b7b9. PMID 23722572
- [Background] Schwab F, Blondel B, Chay E, Demakakos J, Lenke L, Tropiano P, Ames C, Smith JS, Shaffrey CI, Glassman S, Farcy JP, Lafage V. The comprehensive anatomical spinal osteotomy classification. Neurosurgery. 2014 Jan;74(1):112-20; discussion 120. doi: 10.1227/NEU.0000000000000182o. PMID 24356197
- [Background] Toyone T, Shiboi R, Ozawa T, Inada K, Shirahata T, Kamikawa K, Watanabe A, Matsuki K, Ochiai S, Kaiho T, Morikawa Y, Sota K, Yasuchika A, Gen I, Sumihisa O, Ohtori S, Takahashi K, Wada Y. Asymmetrical pedicle subtraction osteotomy for rigid degenerative lumbar kyphoscoliosis. Spine (Phila Pa 1976). 2012 Oct 1;37(21):1847-52. doi: 10.1097/BRS.0b013e31825bf644. PMID 22565386
- [Background] Chan AK, Lau D, Osorio JA, Yue JK, Berven SH, Burch S, Hu SS, Mummaneni PV, Deviren V, Ames CP. Asymmetric Pedicle Subtraction Osteotomy for Adult Spinal Deformity with Coronal Imbalance: Complications, Radiographic and Surgical Outcomes. Oper Neurosurg. 2020 Feb 1;18(2):209-216. doi: 10.1093/ons/opz106. PMID 31214712
- [Background] Buchowski JM, Bridwell KH, Lenke LG, Kuhns CA, Lehman RA Jr, Kim YJ, Stewart D, Baldus C. Neurologic complications of lumbar pedicle subtraction osteotomy: a 10-year assessment. Spine (Phila Pa 1976). 2007 Sep 15;32(20):2245-52. doi: 10.1097/BRS.0b013e31814b2d52. PMID 17873818
- [Background] Wang H, Li W. Multilevel extended posterior column osteotomy plus unilateral cage strutting for degenerative lumbar kyphoscoliosis. Int Orthop. 2020 Jul;44(7):1375-1383. doi: 10.1007/s00264-020-04632-8. Epub 2020 May 21. PMID 32440815
- [Background] Schwab F, Ungar B, Blondel B, Buchowski J, Coe J, Deinlein D, DeWald C, Mehdian H, Shaffrey C, Tribus C, Lafage V. Scoliosis Research Society-Schwab adult spinal deformity classification: a validation study. Spine (Phila Pa 1976). 2012 May 20;37(12):1077-82. doi: 10.1097/BRS.0b013e31823e15e2. PMID 22045006
- [Background] Smith JS, Singh M, Klineberg E, Shaffrey CI, Lafage V, Schwab FJ, Protopsaltis T, Ibrahimi D, Scheer JK, Mundis G Jr, Gupta MC, Hostin R, Deviren V, Kebaish K, Hart R, Burton DC, Bess S, Ames CP; International Spine Study Group. Surgical treatment of pathological loss of lumbar lordosis (flatback) in patients with normal sagittal vertical axis achieves similar clinical improvement as surgical treatment of elevated sagittal vertical axis: clinical article. J Neurosurg Spine. 2014 Aug;21(2):160-70. doi: 10.3171/2014.3.SPINE13580. Epub 2014 Apr 25. PMID 24766290
- [Background] Fei H, Li WS, Sun ZR, Jiang S, Chen ZQ. Effect of patient position on the lordosis and scoliosis of patients with degenerative lumbar scoliosis. Medicine (Baltimore). 2017 Aug;96(32):e7648. doi: 10.1097/MD.0000000000007648. PMID 28796046
- [Background] Han F, Weishi L, Zhuoran S, Qingwei M, Zhongqiang C. Sagittal plane analysis of the spine and pelvis in degenerative lumbar scoliosis. J Orthop Surg (Hong Kong). 2017 Jan;25(1):2309499016684746. doi: 10.1177/2309499016684746. PMID 28139188
- [Background] Xu F, Sun Z, Li W, Hou X, Jiang S, Zhou S, Zou D, Li Z. Correlation between lordosis distribution index, lordosis tilt, and occurrence of proximal junctional kyphosis following surgery for adult degenerative scoliosis. Eur Spine J. 2022 Feb;31(2):267-274. doi: 10.1007/s00586-021-07090-x. Epub 2022 Jan 25. PMID 35075515